CLINICAL TRIAL: NCT03779685
Title: GENe EXpression in Tissues From Operating Field After Regional or General ANesthesia in Patients Undergoing Breast Cancer Surgery. The GENEXAN Randomized Controlled Genomic Trial
Brief Title: GENe EXpression After Regional or General ANesthesia in Patients Undergoing Breast Cancer Surgery
Acronym: GENEXAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Zhirajr Mokini M.D., Principal Investigator, Azienda Ospedaliera San Gerardo di Monza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GENEXAN
Record Dates: First submitted 2018-11-29; First posted 2018-12-19 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): Breast cancer surgery (Tumor Stage 1-3, Nodes 0-2 as determined according to the NCI stage definitions http://www.cancer.gov/cancertopics/pdq/treatment/breast/HealthProfessional/page3/print)
  Interventions: Procedure: General anesthesia
- Regional anesthesia (Experimental): Breast cancer surgery (Tumor Stage 1-3, Nodes 0-2 as determined according to the NCI stage definitions http://www.cancer.gov/cancertopics/pdq/treatment/breast/HealthProfessional/page3/print)
  Interventions: Procedure: Regional anesthesia

INTERVENTIONS:
Procedure: General anesthesia — Sevoflurane and morphine
  Arms: General anesthesia
Procedure: Regional anesthesia — Paravertebral block
  Arms: Regional anesthesia

SUMMARY:
Breast cancer is the most commonly diagnosed cancer in females and the second leading cause of death from cancer in women. It was estimated that 2 million new cases have occurred in 2018 worldwide 1.

Standard anesthetic procedures for the surgery of breast cancer include general and regional anesthesia 2. Growing preclinical and clinical data support the hypothesis that anesthetic choice may affect cancer-related outcomes.

Recurrence in breast cancer was reduced to four-fold in a retrospective study with a 2.5 to 4 year follow up 3. Recurrence and metastasis-free survival, with multivariate analysis, was 94% (95% CI 87,100) versus 82% (74, 91) at 24 months, and 94 (87, 100) versus 77 (68, 87) at 36 months in the paravertebral and general anesthesia patients, respectively, (p=0.013). Currently large confirmatory randomized trials evaluating breast cancer recurrence in patients operated with general or regional anesthesia are yet undergoing 4.

DETAILED DESCRIPTION:
Background: Exposure to general or regional anesthesia, can modulate differently breast cancer biology through a direct activity on cancer cells or indirectly through modifications in host response (immune system, angiogenesis, nervous system). Alterations occur both systemically and locally on the surgical site and is supposed that can affect cancer-related outcomes after months or years.

It is not known whether the action of this short exposure to anesthetics on the host and cancer biology is driven by epigenetic alterations in gene and protein expression during the immediate to early post-anesthesia period.

An altered gene and protein expression profile may affect the response of the immune system, angiogenesis and the nervous system and induce more or less propitious conditions to tumor progression. Data from studies in animals and humans show that gene expression may change in the brain and heart after only a short exposure to general anesthesia and that changes may persist for several weeks.

Methods: The GENEXAN is a randomized, controlled, monocentric, genomic trial aiming to test the hypothesis that regional (paravertebral) anesthesia, compared to general anesthesia, would elicit a differential gene and protein expression pattern in cancer tissue and normal surgical microenvironment after breast cancer surgery in women.

Discussion: This research will serve to map gene and protein expression profile after surgery with different anesthetics and elucidate which genes specific to biological systems may affect tumor biology in the immediate operative period.

The findings may also address further research depending on the tissue specificity of the up or down-regulated genes.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-85 years old
* No undergoing pregnancy
* ASA Score I-IV
* Patients scheduled for breast surgery
* No contraindications (including surgical) to regional (paravertebral) anesthesia
* No previous breast surgery
* No known hereditary or familial cancer syndromes
* No previous cancer anamnesis, radio o chemiotherapy
* Primary breast cancer with Tumor classification 1-3, Nodes 0-2 as determined
* according to the NCI stage definitions (Primary breast cancer without known extension beyond the breast and axillary nodes)
* Free from pain in preoperative period
* Patients who don't use analgesic drugs before surgery
* Patients without cognitive impairment or mental retardation

Exclusion Criteria:

* Women > 18, < 85 years old
* Pregnancy
* ASA Score > IV
* Previous breast surgery
* Contraindications to regional anesthesia
* Known hereditary or familial cancer syndromes
* Previous cancer anamnesis, radio or chemiotherapy
* Tumor classification > 3, Nodes > 2, M > 0 as determined according to the NCI stage
* definitions
* Pain in preoperative period
* Use of analgesic drugs before surgery
* Cognitive impairment or mental retardation
* Patients who did not gave a written informed consent
* Undergoing therapy with alpha (doxazosin) or beta blockers.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Whole genome expression by microarray | before tumor excision
  tumor, biopsy, normal wound tissue
Whole genome expression by mircoarray | during surgery (just after tumor excision)
  tumor, wound tissue

SECONDARY OUTCOMES:
Immune progenitors (MDBCs, GMPs, HPSCs), Natural Killer, T regulatory Lymphocytes, PentraxinIII | before tumor excision
  in blood
cancer recurrence | each 6 months for up to 7 years
  local or distant metastasis
survival from cancer | each 6 months for up to 7 years
  death
Immune progenitors (MDBCs, GMPs, HPSCs), Natural Killer, T regulatory Lymphocytes, PentraxinIII | at the end of surgery
  in blood
Immune progenitors (MDBCs, GMPs, HPSCs), Natural Killer, T regulatory Lymphocytes, PentraxinIII | at 24 hours
  in blood
Immune progenitors (MDBCs, GMPs, HPSCs), Natural Killer, T regulatory Lymphocytes, PentraxinIII | at 168 hours
  in blood

IPD SHARING:
Plan to Share IPD: No